CLINICAL TRIAL: NCT04077983
Title: a Single-arm Study of Nab-Paclitaxel Combined With Gemcitabine Adjuvant Chemotherapy After Radical Resection of Intrahepatic Cholangiocarcinoma
Brief Title: Nab-Paclitaxel Combined With Gemcitabine Adjuvant Chemotherapy After Radical Resection of Intrahepatic Cholangiocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ICC-afterresection
Record Dates: First submitted 2019-09-01; First posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Cholangiocarcinoma, Intrahepatic
Keywords: intrahepatic cholangiocarcinoma; nab-paclitaxel and gemcitabine chemotherapy
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combined therapy using nab-paclitaxel and gemcitabine chemo (Experimental): 1. Day1 nab-paclitaxel 125mg/m2, Day8 nab-paclitaxel 125mg/m2
  2. Day1 gemcitabine 1000mg/m2, Day8 gemcitabine 1000mg/m2
  3. Three weeks is a course of treatment with a total of 4 courses.
  Interventions: Drug: combined therapy using nab-paclitaxel and gemcitabine chemotherapy

INTERVENTIONS:
Drug: combined therapy using nab-paclitaxel and gemcitabine chemotherapy — 1. Day1 nab-paclitaxel 125mg/m2, Day8 nab-paclitaxel 125mg/m2
  2. Day1 gemcitabine 1000mg/m2, Day8 gemcitabine 1000mg/m2
  3. Three weeks is a course of treatment with a total of 4 courses.

SUMMARY:
In this phase 2 study, we aim to evaluate the effects and safety of combined therapy using nab-paclitaxel and gemcitabine chemotherapy for patients after radical resection of Intrahepatic Cholangiocarcinoma

DETAILED DESCRIPTION:
Most patients with intrahepatic cholangiocarcinoma (ICC) are often accompanied by local or distant metastases and lose the opportunity for surgical resection. Surgical resection is the only effective means for long-term survival of patients with intrahepatic cholangiocarcinoma. However, multiple tumors, lymph node metastasis, and vascular invasion significantly reduced postoperative survival. Most patients will relapse due to less clinical data. The best adjuvant treatment strategy and standard protocol for patients with intrahepatic cholangiocarcinoma has not been determined. Current treatment options include chemotherapy based on fluoropyrimidine or gemcitabine. Albumin-bound paclitaxel(nab-paclitaxel) has been used to treat a variety of malignancies such as non-small cell lung cancer, pancreatic cancer, breast cancer, melanoma, ovarian cancer and the like. In the field of pancreatic cancer, studies have confirmed that albumin-bound paclitaxel has synergistic effects with gemcitabine. The combination of gemcitabine alone significantly increased the intratumoral concentration of gemcitabine. Albumin-bound paclitaxel plus gemcitabine is the first choice for first-line treatment of pancreatic cancer, but clinical studies in the field of cholangiocarcinoma are very limited. Based on the same origin of pancreatic and biliary embryos, biological behavior and pathological similarities. Therefore, in this second phase of the study, our aim was to evaluate the efficacy and safety of chemotherapy with nab-paclitaxel and gemcitabine in the prevention of postoperative recurrence in patients with intrahepatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must have good compliance, be understood the research process of this study and required to sign an informed consent form;
2. age 18-75 years old, male or female;
3. Histopathologically confirmed intrahepatic cholangiocarcinoma，excluding mixed liver cancer;
4. The longest diameter of a single tumor in patients before surgery is 3~9cm. If the number of multiple tumors is ≤3, the total diameter≤9cm, maximum diameter ≤5cm;
5. Study treatment can be started within 4~6 weeks after R0 resection;
6. Except for R0 resection, no other anti-tumor treatment has been received;
7. No distant transfer；
8. ECOG<2, or KPS>70；
9. Bone marrow function criteria: hemoglobin (HGB)≥90g/L; absolute neutrophil count (ANC)≥1.5×109/L; platelets (PLT)≥100×109/L;
10. Liver function criteria: ALT, AST≤5×ULN, serum total bilirubin<3×ULN;
11. Renal function criteria: creatinine clearance > 45 mL/min
12. Prothrombin time <14s; (no anticoagulant therapy);
13. Patients without biliary obstruction who require biliary stent implantation must be completed at least 7 days prior to enrollment;
14. Non-lactating or pregnant women, contraception during or after 6 months of treatment.
15. No contraindications for gemcitabine and Nab-paclitaxel.

Exclusion Criteria:

1. Those patients who are allergic to the chemotherapy drugs and their components in this study
2. Patients with other malignant tumors within 5 years (except for cured carcinoma in situ or basal cell carcinoma of the skin)
3. Concomitant diseases that may interfere with treatment studies: such as severe infections, HIV-positive, clinically severe (ie active) Heart disease, uncontrolled epilepsy, central nervous system disease, or history of mental disorders;
4. Intraoperative or postoperative pathology determines patients who do not meet radical resection;
5. Patients with current or previous ≥ grade II peripheral neuropathy;
6. Patients who participated in other clinical studies within 4 weeks prior to enrollment;
7. Patients who has undergone organ transplantation;
8. Patients considered by the investigator not suitable for this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 24 months
  the time from the day after surgery to the recurrence of cancer.

SECONDARY OUTCOMES:
safety: the potential side effects | 6 months
  the potential side effects

OTHER OUTCOMES:
overall survival | 24 months
  the time from the day after surgery to death

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, MD&PhD, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Desai N, Trieu V, Yao Z, Louie L, Ci S, Yang A, Tao C, De T, Beals B, Dykes D, Noker P, Yao R, Labao E, Hawkins M, Soon-Shiong P. Increased antitumor activity, intratumor paclitaxel concentrations, and endothelial cell transport of cremophor-free, albumin-bound paclitaxel, ABI-007, compared with cremophor-based paclitaxel. Clin Cancer Res. 2006 Feb 15;12(4):1317-24. doi: 10.1158/1078-0432.CCR-05-1634. PMID 16489089
- [Background] Frese KK, Neesse A, Cook N, Bapiro TE, Lolkema MP, Jodrell DI, Tuveson DA. nab-Paclitaxel potentiates gemcitabine activity by reducing cytidine deaminase levels in a mouse model of pancreatic cancer. Cancer Discov. 2012 Mar;2(3):260-269. doi: 10.1158/2159-8290.CD-11-0242. Epub 2012 Feb 28. PMID 22585996
- [Background] Von Hoff DD, Ramanathan RK, Borad MJ, Laheru DA, Smith LS, Wood TE, Korn RL, Desai N, Trieu V, Iglesias JL, Zhang H, Soon-Shiong P, Shi T, Rajeshkumar NV, Maitra A, Hidalgo M. Gemcitabine plus nab-paclitaxel is an active regimen in patients with advanced pancreatic cancer: a phase I/II trial. J Clin Oncol. 2011 Dec 1;29(34):4548-54. doi: 10.1200/JCO.2011.36.5742. Epub 2011 Oct 3. PMID 21969517